CLINICAL TRIAL: NCT05682976
Title: Prospective Multicentre Study on Ophthalmological Adverse Events of Tralokinumab in the Treatment of Atopic Dermatitis
Brief Title: Ophthalmological Adverse Events of Tralokinumab in AD
Acronym: TRALO-Oeil
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: RC22_0628
Record Dates: First submitted 2022-12-09; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis, Tralokinumab, adverse event, conjunctivitis
MeSH Terms: conditions — Dermatitis, Atopic; Conjunctivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AD patient treated by Tralokinumab: AD patient treated by Tralokinumab

SUMMARY:
Atopic dermatitis (AD) is a skin disease characterised by xerosis, pruritus and erythematous plaques. It is common in children (10 to 20%) with an increasing prevalence (multiplied by 2 in 20 years) and begins to develop at 3 months of age. Half of all atopic dermatitis cases disappear by the age of 5, but 10 to 15% of cases persist into adulthood (i.e. about 3.5% of the French adult population). Conventional treatments consist of emollient creams, topical corticosteroid, topical immunomodulators (topical calcineurin inhibitor: tacrolimus) or systemic cyclosporine. However, a proportion of patients (10%) do not respond sufficiently to this therapeutic arsenal. Recent therapies using monoclonal antibodies (biotherapies) are available (DUPILUMAB -anti Interleukin-4 (IL4) antibody and soon TRALOKINUMAB-anti Interleukin-L13 (IL13) antibody). Conjunctivitis is an adverse event reported in patients treated with dupilumab and tralokinumab in clinical trials. Given that baseline ophthalmic comorbidities affect approximately 20% of AD patients, it is crucial to include an evaluation in future prospective real-life longitudinal studies to assess the true incidence of biologic-induced ophthalmic adverse events. No such study is currently available for Tralokinumab. The French group GREAT (GROUPE DE RECHERCHE SUR L'ECZEMA ATOPIQUE) has recently conducted a study on ocular adverse events of dupilumab (DUPI-ŒIL study, I. COSTEDOAT, M. WALLAERT et al, submitted) which included 180 patients followed for at least 4 months. The results show that the majority of dupilumab-induced conjunctivitis is de novo (frequency 18%). Conjunctivitis-type adverse events were also reported at a frequency of 3.0% to 11.0% in the ECZTRA pivotal studies with Tralokinumab. However, the ophthalmological impact of IL13 inhibition remains partially unknown. Further characterisation of ophthalmological adverse events in patients treated with Tralokinumab in real life is needed to provide information for future recommendations (including prioritisation of indications for systemic therapy) and to improve compliance. The primary objective of the TRALO-OEIL study is to determine the frequency of occurrence of ophthalmologic adverse events with TRALOKINUMAB.

DETAILED DESCRIPTION:
The study consists of following over 12 months patients who have been prescribed Tralokinumab to treat their AD.

The inclusion visit takes place on the day of initiation of TRALOKINUMAB. Current ophthalmic follow-up recommendations include an initial examination before the start of treatment and then regularly during treatment and in case of ocular events. Patients are advised to consult the ophthalmology department of the university hospital where they are treated promptly in case of ophthalmological adverse events.

The investigators will collect data from the initial routine visit (M0) and from visits at 4 months (M4) and 12 months (M12).

Any other visits for ocular events during follow-up will be collected (Unscheduled visits).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years),
* Patients with atopic dermatitis,
* Patients indicated for treatment with Tralokinumab
* Patients able to express non opposition.

Exclusion Criteria:

* Patients who have stopped Dupilumab for less than one month,
* Patients under guardianship or trusteeship
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for AD requiring systemic treatment with Tralokinumab. In order to keep a representative overview of all patients with atopic dermatitis, the number of patients included after Dupilumab failure will be limited to 25%.
  For patients previously treated with Dupilumab, a washout period of up to one month should be observed prior to inclusion to avoid the reporting of ophthalmological events at baseline still related to Dupilumab treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
occurrence of an ophthalmologic adverse event (conjunctivitis, keratoconjunctivitis, etc.) | 4 months
  the occurrence of an ophthalmologic adverse event (conjunctivitis, keratoconjunctivitis, etc.) 4 months after initiation of treatment with TRALOKINUMAB or an increase in a pre-existing ophthalmologic condition on treatment

SECONDARY OUTCOMES:
Occurrence or worsening of conjunctivitis, keratoconjunctivitis, blepharitis | 4 months
  Occurrence or worsening of conjunctivitis, keratoconjunctivitis, blepharitis,... within 4 months of initiation of TRALOKINUMAB
Occurrence or worsening of conjunctivitis, keratoconjunctivitis, blepharitis | 12 months
  Occurrence or worsening of conjunctivitis, keratoconjunctivitis, blepharitis,... within 12 months of initiation of TRALOKINUMAB
Severity score of ophthalmological damage | 12 months
  Severity score of ophthalmological damage used in a previous study (DUPI-ŒIL study, I. Costedoat, M. Wallaert et al, submitted). minimum value: 0, maximum value: 68. A lower score mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien BARBAROT, PHPH, Principal Investigator — Nantes University Hospital
Locations (11):
- France (11):
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHu de Dijon, Dijon
  - CHRU de Lille, Lille
  - Hospice Civil de Lyon, Lyon
  - CHU de Nantes, Nantes
  - Hôpital Saint Louis, Paris
  - CHu de Poitiers, Poitiers
  - CHu de Rennes, Rennes
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: Undecided